CLINICAL TRIAL: NCT03212378
Title: Safety and Efficacy of "Standardized" Complex High-risk Interventional Procedures - a New Pathway for Protected Percutaneous Coronary Interventions
Brief Title: Safety and Efficacy of "Standardized" CHIP
Status: Completed | Type: Observational
Sponsor: University Hospital, Essen (Other)
Responsible Party: Principal Investigator, Fadi Al-Rashid, Principal Investigator, University Hospital, Essen
Other Study IDs: FA_2017_01
Record Dates: First submitted 2017-07-03; First posted 2017-07-11 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- CHIP 1 - low risk patients
  Interventions: Other: percutaneous coronary interventions
- CHIP 2 - medium risk patients
  Interventions: Other: percutaneous coronary interventions
- CHIP 3 - high risk patients
  Interventions: Other: percutaneous coronary interventions

INTERVENTIONS:
Other: percutaneous coronary interventions — Percutaneous coronary intervention.

SUMMARY:
In routine clinical practice, high-risk patients with high-risk anatomies are more often referred for interventional treatment by percutaneous coronary interventions (PCI). Current guidelines only suggest that elective insertion of an appropriate hemodynamic support device as an adjunct to PCI may be reasonable in selected high-risk patients.

The objective of this study is to investigate the safety and efficacy of a "standardized program" for complex high-risk interventional procedures (CHIP).

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent
* Non emergent PCI of at least one de novo or restenotic lesion in a native coronary vessel or bypass graft

Exclusion Criteria:

* Subject has uncorrectable abnormal coagulation parameters (defined as platelet count ≤75,000/mm3 or INR ≥2.5.)
* History of recent (within 1 month) stroke or TIA
* Allergy or intolerance to heparin, aspirin, ADP receptor inhibitors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of consecutive high-risk subjects indicated for percutaneous complex high-risk interventional procedures.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2016-01-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Safety & feasibility | 30 days
  Accurate classification of patients into the respective group defined by the necessity of upgrade
Hemodynamic Compromise (HC) | 30 days.
  Freedom from hemodynamic compromise during PCI procedure defined as: mean arterial pressure (MAP) not decreasing to values below 60 mmHg for more than 10 minutes during the PCI procedure

SECONDARY OUTCOMES:
Major Adverse Cardiac and Cerebrovascular Events (MACCE) | 30 days
  A composite rate of the following intra-procedural and post-procedural Major Adverse Cardiac and Cerebrovascular Events (MACCE) events defined as death, new myocardial infarction, or cerebrovascular accident up to 30 days post index procedure.
Adverse events | 30 days
  Rates of acute kidney injury ([AKI] according to KDIGO), sepsis, vascular complications (defined by Valve Academic Research Consortium 2 [VARC 2]), bleeding (defined by Bleeding Academic Research Consortium [BARC]) and coronary complications.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Essen, Essen, North Rhine-Westphalia, Germany